CLINICAL TRIAL: NCT06288152
Title: Evaluation of Thiosulfate Enhanced Organ Preservation Solution in Kidney Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alp Sener (Other)
Responsible Party: Sponsor-Investigator, Alp Sener, Alp Sener MD PhD FRCSC Lavergne Chair and Professor of Urology City-wide Head of Urology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STS-Transplant
Record Dates: First submitted 2024-01-16; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Renal Transplant; Kidney Transplant
Keywords: Thiosulfate; Transplant; Renal; Kidney
MeSH Terms: interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): STS plus standard of care
  Interventions: Drug: Sodium Thiosulfate
- Control Group (No Intervention): Standard of care

INTERVENTIONS:
Drug: Sodium Thiosulfate — 0.15 mL administered
  Other Names: Seacalphyx
  Arms: Intervention Group

SUMMARY:
End-stage renal disease (ESRD) is a significant clinical problem for which dialysis or transplantation is required. The current need for kidneys for transplantation vastly exceeds the supply available from live donors, necessitating the use of kidneys from deceased donors. However, kidneys from deceased donors are associated with reduced viability, as lack of blood supply upon cardiac death increases tissue damage. In addition, the standard protocol for cold preservation of donor kidneys between procurement and transplantation increases the risk of delayed donor kidney function by 23% for every 6-hours of storage. Moreover, compared to other organs, the kidney is particularly prone to transplantation-induced injury due to its high metabolic activities and oxygen consumption. Hence, any minor disturbances in blood supply can easily lead to kidney injury. Therefore, it is not surprising that deceased donor kidneys have a low tolerance for damage associated with lack of blood supply. The focus of the investigators research has been to pioneer the development and supplementation of existing kidney preservation solutions with novel hydrogen sulfide (H2S) donor molecules to improve kidney viability for clinical transplantation. Specifically, the investigators demonstrated that supplementation of standard kidney preservation solutions with non-clinically viable H2S donor molecules significantly increased donor kidney protection and prolonged transplant recipient survival in murine and porcine models of kidney transplantation. Having shown the same salutary effect using sodium thiosulfate (STS; a clinically viable H2S donor drug) in rat kidney transplantation, the investigators aim to repeat this work using STS in porcine and clinical kidney transplantation.

This single-blind study will enroll participants receiving a kidney transplant. Through randomization, half of the participants will receive STS through administration into the pump the kidney is placed on after procurement from the donor and before transplant to the recipient. Participants will be followed for 1-year post transplant where blood and urine will be collected to determine graft function.

DETAILED DESCRIPTION:
Full description pending

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* End-Stage Renal Disease
* Receiving a kidney transplant from a deceased donor (NDD or DCD)

Exclusion Criteria:

* Under 18 years of age
* Inability to provide informed consent
* Living donor kidney recipients
* Pregnant individuals
* Known allergy to study medication or its components (non-medicinal ingredients)
* Multiorgan transplant patients such as simultaneous kidney pancreas or liver kidney transplants
* Currently enrolled in another interventional transplant clinical trial, or another clinical trial that in the opinion of the QI and PI would greatly impact the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Effects of STS will be measured by: Delayed graft function | 1 year
  Number of participants requiring dialysis use post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Alp Sener, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
Study report
Supporting Information: CSR
Time Frame: After study completion
Access Criteria: To be determined